CLINICAL TRIAL: NCT04842890
Title: Phase II Study of Pencil Beam Scanning Proton Stereotactic Body Radiation Therapy for Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The New York Proton Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYPC ERC# 2020-027
Record Dates: First submitted 2021-03-15; First posted 2021-04-13 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Stereotactic body radiation therapy (SBRT) with Pencil Beam Scanning (PBS) proton therapy (Other)
  Interventions: Radiation: Pencil Beam Scanning Proton SBRT

INTERVENTIONS:
Radiation: Pencil Beam Scanning Proton SBRT — The intervention being investigated is ultra-hypofractionated, image-guided, pencil beam scanning proton SBRT directed at the prostate gland and seminal vesicles to 40 Gy equivalent in 5 fractions, delivered every other day.

SUMMARY:
This is a single arm phase II study of image-guided pencil beam scanning proton SBRT (40Gy RBE in 5 fractions delivered every other day) for patients with low- and intermediate-risk prostate cancer. The primary aim is to assess GU/GI toxicity of proton SBRT and compare this to historic outcomes associated with photon-based prostate SBRT. The primary endpoint is 2-year grade 3+ GU/GI toxicity free rate by CTCAE v5.0, which is expected to be ≥95%. Toxicity will be evaluated by the treating radiation oncologist at least once during SBRT, then following SBRT at 1, 3, 6, 12, 18, and 24 months. The treatment will be considered safe if grade 3 or higher GU/GI toxicity free rate at 2 years is >85% (95% rate expected with a 10% non-inferiority margin). The accrual goal is 61 patients over 3 years. To ensure that unexpected significant toxicity is identified, all grade 3 or higher toxicities will be reported to the study PI and the trial will stop accruing if at any point 4 or more patients experience a grade 3 or higher toxicity after completing SBRT. This is felt to be conservative given the vast experience with photon SBRT at this dose with an expected G3+ toxicity of ~5%.

Secondary objectives are to examine patient-reported urinary, gastrointestinal, sexual, and financial outcomes using IPSS, EPIC-26, and COST questionnaires at the same follow-up timepoints as above. Baseline measures of these domains will be obtained prior to treatment as well. Clinical outcomes will also be evaluated with PSA measured at each follow-up, as well as prostate MRI and biopsies at 2 years. Patients will be followed for at least 2 years to determine rates of PSA relapse, salvage treatment, development of metastases, death from prostate cancer, and overall survival. A dosimetric comparison will be performed where each patient will be planned for proton and photon SBRT to determine possible advantages of proton SBRT.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven NCCN low- or intermediate-risk prostate cancer, which includes patients with:
* Gleason score ≤7 disease
* PSA ≤20 ng/ml
* Clinical T1-T2c disease

  * Note: Patients who only have radiographic evidence of possible or probable T3 disease (i.e., extracapsular extension or seminal vesical invasion) will not be excluded.
* KPS ≥ 80%
* Prostate size as determined on MRI to be < 100 cc. Prostate size can be determined on CT scan if MRI is not available.
* Male 18 years of age or older
* IPSS ≤ 20
* Patient must be a candidate for and agree to placement of intraprostatic fiducial markers and a hydrogel rectal spacer
* Patient must be available for at least 2 years of follow-up

Exclusion Criteria:

* Prior prostate surgery (including cryosurgery)

  * Note: Patients who underwent TURP or greenlight PVP are eligible if it was > 12 weeks prior to the anticipated start date of SBRT
* Prior history of chronic prostatitis or urethral stricture
* Currently active cancer(s) other than non-melanoma skin cancers. Patients are not considered to have currently active cancers if they have completed therapy and are considered by their physicians to be at <5% risk of relapse within 2 years.
* Life expectancy of < 2 years

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 61 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
1. Grade 3+ GU/GI toxicity-free rate determined by CTCAE v5.0 grading. | 2 years
  The NCI Common Terminology Criteria for Adverse Events v5.0 is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term.

SECONDARY OUTCOMES:
1. Patient reported urinary symptoms determined by IPSS. | 2 years
  The International Prostate Symptom Score (IPSS) was developed to assess the severity of lower urinary tract symptoms associated to Benign Prostatic Hyperplasia and has also been applied to other conditions that cause LUTS. The IPSS consists of a total of seven questions that deal with voiding symptoms (incomplete empty, intermittency, weak stream and straining to void) and storage symptoms (frequency, urgency and nocturia) and an additional question to measure quality of life. The score ranges from 0 to 35, with lower scores denoting a better health state.
2. Patient reported urinary, bowel, and hormonal quality of life determined by EPIC-26. | 2 years
  EPIC-26 is the "Expanded Prostate Cancer Index Composite" patient reported outcomes questionnaire. A clinical tool to assess urinary, bowel, sexual and vitality health. The score from each of the 5 domains runs from 0 (none) to 12 (severe) impact on quality of life. Each domain score when added together gives an overall score of zero (unaffected) to 60 (severely affected)
3. Patient reported financial toxicity determined by COST | 2 years
  Comprehensive Score for Financial Toxicity Functional Assessment of Chronic Illness Therapy (COST-FACIT) was developed as part of a series of questionnaires aimed at measuring different symptom indexes of health-related quality of life in patients with advance disease such as cancer. The survey contains 12 questions and each of them is rated from 0 (not at all) to 4 (very much). This survey focuses on financial distress caused by illness in patients with cancer. It takes about 5 minutes to complete.
4. 2-year and 5-year biochemical progression free survival | 2 years and 5 years
  Biochemical failure is defined as a sustained rise in PSA of 2 ng/mL or more above the nadir (the lowest PSA level after radiotherapy).
5. 2-year local control determined by MRI and biopsies | 2 years
6. 2-year and 5-year metastasis free survival | 2 years and 5 years
7. 2-year and 5-year prostate cancer specific survival | 2 years and 5 years
8. 2-year and 5-year overall survival | 2 years and 5 years
9. Dosimetric advantages determined by target coverage, conformality, and normal tissue sparing | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Gorovets, MD, Principal Investigator — The New York Proton Center; Shaakir Hasan, DO, Principal Investigator — The New York Proton Center
Locations (1):
- The New York Proton Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided